CLINICAL TRIAL: NCT06032195
Title: A Prospective Randomized Single Blind Multicenter Phase II Study of Organ Perfusion With Custodiol-N Compared With Custodiol in Heart Transplantation in Children
Brief Title: Study of Organ Perfusion in Heart Transplantation in Children
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. F. Köhler Chemie GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CL-N-HTX-Paed-II/10/20
Record Dates: First submitted 2023-08-21; First posted 2023-09-11 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Heart Transplantation
MeSH Terms: interventions — Custodiol-N solution; Solutions; Organ Preservation; Transplantation

STUDY DESIGN:
Who Masked: Participant
Masking Description: The patient and their legal representatives will be blinded to treatment. All other parties are unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Custodiol-N (Experimental): organ will be perfused with Custodiol-N solution
  Interventions: Drug: Custodiol-N
- Custodiol (Active Comparator): organ will be perfused with Custodiol solution
  Interventions: Drug: Custodiol

INTERVENTIONS:
Drug: Custodiol-N — heart will preserved in and will be treated with Custodiol-N solution
  Other Names: Solution for organ preservation in transplantation
  Arms: Custodiol-N
Drug: Custodiol — heart will preserved in and will be treated with Custodiol solution
  Other Names: Solution for organ preservation in transplantation
  Arms: Custodiol

SUMMARY:
The goal of this prospective randomized single blind multicenter phase II study is to compare organ perfusion with Custodiol-N and Custodiol in heart transplantation in children of all ages (birth to <18 years) being listed on the waiting list for heart transplantation. The main question it aims to answer is:

to compare the safety of Custodiol-N in heart transplantation in children in comparison to its precursor product Custodiol.

Participants will receive either a heart to be transplanted, either perfused with Custodiol-N or Custodiol to Researchers will compare the two solutions to see if the new solution Custodiol-N is safe in heart transplantation in children.

DETAILED DESCRIPTION:
Orthotopic Heart transplantation (or cardiac transplantation) is a procedure performed in patients with end stage heart failure when other treatments have failed.

The surgical procedures for orthotopic heart transplantation are essentially the same in adult and paediatric patients . Due to anatomical variants in congenital heart disease the procurement procedure may be modified with regard to the extent of the Vena cava superior and the great vessels. In implantation most frequently the bicaval technique is used but the biatrial technique which is leaving the back wall of both atria in situ may also be employed.

A main difference between adult and paediatric heart transplantation (HTx) are the indications for transplantation: In adults the majority of patients undergo HTx as treatment of end stage heart failure due to cardiomyopathy or severe coronary artery disease when other treatments have failed. Infants younger than one year of age congenital heart disease (CHD) is the most common diagnosis representing more than every second case followed by dilated cardiomyopathy (DCM) in more than one third of cases. In older patients DCM is the most frequent underlying diagnosis. CHD may include patients who have undergone corrective surgery and in whom myocardial dysfunction develops later .

ELIGIBILITY:
Inclusion Criteria:

* Age from birth to less than18 years
* Recipients awaiting their first transplant
* Ability of the patients and/ or their legal guardians to understand character and individual consequences of the clinical trial
* written informed consent of the patients and/ or their legal guardians (must be available before enrolment in the study)
* Patient listed on the waiting list for heart transplantation

Exclusion Criteria:

* Patients who have participated within 30 days or are still participating in any other interventional studies
* history of severe organic disease other than concerning the heart
* history/demonstration of HIV antibodies or AIDS
* multiorgan transplantation
* machine-perfused organ
* the explantation team is affiliated to another clinic than transplantation team
* Failing Fontan patients
* Patients who have been incarcerated or involuntarily institutionalized by court order or by the authorities
* Pregnancy and lactation

Ages: 24 Hours to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
adverse event reporting | up to 3 months
  Safety assessment

SECONDARY OUTCOMES:
heart rate | up to day 7 after release of the aortic cross clamp
  vital parameters
blood pressure (systolic (SBP) and diastolic (DBP)) | up to day 7 after release of the aortic cross clamp
  vital parameters
body temperature | up to day 7 after release of the aortic cross clamp
  vital parameters
concentration of cardiac troponin | up to day 7 after release of the aortic cross clamp
  laboratory tests
concentration of creatinine kinase (CK-MB) | up to day 7 after release of the aortic cross clamp
  laboratory tests
(SBP (systolic blood pressure), DBP (diastolic blood pressure)) | from termination of cardiopulmonary bypass until transfer to intensive care unit
  Haemodynamics
Heart Rhythm (HR) | from termination of cardiopulmonary bypass until transfer to intensive care unit
  Haemodynamics
Pulmonary artery pressure (PAP (if available)) | from termination of cardiopulmonary bypass until transfer to intensive care unit
  Haemodynamics
Cerebrovascular resistance (CVP (if available)) | from termination of cardiopulmonary bypass until transfer to intensive care unit
  Haemodynamics
Death | up to 12 months
  survival
function of transplanted organ (heart) | up to 12 months
  Graft survival
Readmission to intensive care unit (ICU) | up to 12 months
  return to intensive care unit
Length of ICU stays | up to 12 months
  duration of stay in intensive care unit
Catecholamine requirement | up to day 7
  (yes/no)
Antihypertensives intake | up to 12 months
  (yes/no)
Milrinone support | up to day 7
  (yes/no)
Need for pacemaker therapy | up to day 7
  (yes/no)
Left and right ventricular assist device (LVAD, RVAD) | up to 12 months
  Device therapy (each yes/no)
Extracorporeal membrane oxygenation (ECMO) | up to 12 months
  Device therapy (each yes/no)
Biventricular assist Device (BIVAD) or percutaneous LVAD | up to 12 months
  Device therapy (each yes/no)
Ejection fraction | up to day 7
  Echocardiographic markers of function and rejection
enddiastolic and endsystolic ventricle | up to day 7
  Echocardiographic markers of function and rejection
Cardiac arrhythmias | up to day 7
  occurrence, severity, type

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Knosalla, Prof. Dr., Principal Investigator — Deutsches Herzzentrum der Charité
Locations (3):
- Germany (3):
  - Deutsches Herzzentrum der Charité, Berlin
  - Universitätsklinikum Gießen (UKGM), Kinderherzzentrum, Klinikum für Kinderherzchirurgie, Giessen
  - Klinikum der Universität München (LMU), Klinik und Poliklinik für Herzchirurgie, Chirurgische Klinik, München

IPD SHARING:
Plan to Share IPD: No